CLINICAL TRIAL: NCT00645086
Title: A Phase III Comparative Efficacy Study of 5 Days of M02-472 Clarithromycin Extended-Release Tablets to 7 Days of Clarithromycin Immediate-Release Tablets for the Treatment of Subjects With Acute Bacterial Exacerbation of Chronic Bronchitis.
Brief Title: Comparative Study of 5 Days of M02-472 Clarithromycin Extended-Release Tablets to 7 Days of Clarithromycin Immediate-Release Tablets for the Treatment of Exacerbation of Chronic Bronchitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Angela M Nilius, Ph.D., Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-472
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Acute Bacterial Exacerbation of Chronic Bronchitis (ABECB).
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: clarithromycin extended-release tablets
- B (Active Comparator)
  Interventions: Drug: clarithromycin immediate-release tablets

INTERVENTIONS:
Drug: clarithromycin extended-release tablets — 5-day course of clarithromycin extended-release tablets (2 x 500 mg QD)
  Other Names: ABT-268; Biaxin; clarithromycin
  Arms: A
Drug: clarithromycin immediate-release tablets — 7-day course of clarithromycin immediate-release tablets (1 x 500 mg BID)
  Other Names: ABT-268; Biaxin; clarithromycin
  Arms: B

SUMMARY:
To compare the efficacy of a 5-day course of clarithromycin extended-release tablets (2 x 500 mg QD) with that of a 7-day course of clarithromycin immediate-release tablets (1 x 500 mg BID) in the treatment of acute bacterial exacerbation of chronic bronchitis.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory subject who does not require intravenous antibiotic therapy.
* Subject who has a medical history of chronic bronchitis.
* A history of regular medication use (>=3 consecutive months within the past 2 years) to treat pulmonary disease.
* Subject must have evidence of pulmonary function test abnormalities.
* The onset of signs and symptoms of the current exacerbation must occur within 14 days before Evaluation 1.

Exclusion Criteria:

* Medical history of hypersensitivity, allergic or adverse reactions to clarithromycin, erythromycin, or any of the macrolide antibiotics.
* A female who is pregnant or is lactating.
* Subject who has suspected or known (positive chest radiograph) pneumonia.
* Subject who has evidence of significant bronchiectasis (by CT) or atelectasis, active tuberculosis or other mycobacterial infection, bullous emphysema, pulmonary embolism, lung abscess, tumor (primary or metastatic) involving the lung, pleural effusion, or cystic fibrosis that could confound the assessment of signs and symptoms of ABECB.
* Subject who requires parenteral antibiotic therapy.
* Subject who requires hospitalization for treatment of current episode of ABECB.
* Subject who has any other infection or condition, which necessitates use of a concomitant systemic antibiotic.
* Subject who has any underlying condition/disease, which would be likely to interfere with the completion of the course or absorption of study drug therapy or follow-up.
* Subject who has a severe or complicated lower respiratory tract infection or a severely compromised respiratory status (i.e., oxygen dependent, requiring hospitalization).
* Known significant renal or hepatic impairment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2002-12; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Clinical Response | 23 days
Bacteriologic Response | 23 days

SECONDARY OUTCOMES:
Adverse events assessment | 42 days with follow-up to a satisfactory conclusion
Physical exam; Vital signs; Use of other medications and supplements | 42 days
Laboratory evaluations | 23 days

CONTACTS AND LOCATIONS:
Locations (136):
- United States (125):
  - Birmingham, Alabama
  - Columbiana, Alabama
  - Hoover, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Ozark, Alabama
  - Glendale, Arizona
  - Phoenix, Arizona
  - Sun City West, Arizona
  - Tucson, Arizona
  - Camden, Arkansas
  - Clovis, California
  - Corona, California
  - Fountain View, California
  - Fresno, California
  - Huntington Beach, California
  - Lakewood, California
  - Pasadena, California
  - Rancho Cucamonga, California
  - Roseville, California
  - San Diego, California
  - San Jose, California
  - Sylmar, California
  - Temecula, California
  - Torrance, California
  - Upland, California
  - Colorado Springs, Colorado
  - Loveland, Colorado
  - Wheat Ridge, Colorado
  - Waterbury, Connecticut
  - Brandon, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Gainesville, Florida
  - Largo, Florida
  - Merritt Island, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - Panama City, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Blue Ridge, Georgia
  - Fort Gordon, Georgia
  - Marietta, Georgia
  - Rome, Georgia
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Hines, Illinois
  - Orland Park, Illinois
  - Elkhart, Indiana
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Lexington, Kentucky
  - Murray, Kentucky
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Sunset, Louisiana
  - Auburn, Maine
  - Chester, Maryland
  - DeWitt, Michigan
  - Livonia, Michigan
  - Saginaw, Michigan
  - Saint Joseph, Michigan
  - Chesterfield, Missouri
  - Jefferson City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Blackwood, New Jersey
  - Mount Laurel, New Jersey
  - Toms River, New Jersey
  - West Caldwell, New Jersey
  - Astoria, New York
  - Bronxville, New York
  - Buffalo, New York
  - Camillus, New York
  - New York, New York
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Chardon, Ohio
  - Mogadore, Ohio
  - Toledo, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Lake Oswego, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Bensalem, Pennsylvania
  - Fleetwood, Pennsylvania
  - Philadelphia, Pennsylvania
  - Ridley Park, Pennsylvania
  - Cranston, Rhode Island
  - East Providence, Rhode Island
  - Bamberg, South Carolina
  - Greer, South Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Chattanooga, Tennessee
  - Clarksville, Tennessee
  - Ducktown, Tennessee
  - Johnson City, Tennessee
  - New Tazewell, Tennessee
  - Savannah, Tennessee
  - Selmer, Tennessee
  - Austin, Texas
  - Beaumont, Texas
  - Colleyville, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Christianburg, Virginia
  - Mechanicsville, Virginia
  - Newport News, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - Milwaukee, Wisconsin
  - New Berlin, Wisconsin
- Canada (10):
  - Coquitlam, British Columbia
  - Winnipeg, Manitoba
  - Kitchener, Ontario
  - Markham, Ontario
  - Mississauga, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Sherbrooke, Quebec
  - Ste-Foy, Quebec
  - Saskatoon, Saskatchewan
- San Juan, Puerto Rico